CLINICAL TRIAL: NCT07281443
Title: Mass Drug Administration and Targeted Control Against Carriage to Reduce Plasmodium Transmission in the Sahel - Administration de Masse d'Antipaludiques et Lutte ciblée Contre le Portage Pour REduire la Transmission de Plasmodium au Sahel
Brief Title: MDA and Targeted Control Against Plasmodium Carriage in the Sahel
Acronym: AMARETI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Programme National de Lutte contre le Paludisme (PNLP), Senegal (Unknown); L'université de Thiès (Other); Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024_SESSTIM_AMARETI; 23SANIC216 (Other Grant/Funding Number: L'Initiative/Expertise France); ANR-23-CE35-0002 (Other Grant/Funding Number: Agence Nationale de la Recherche)
Record Dates: First submitted 2025-09-29; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Malaria, Falciparum; Malaria, Asymptomatic Parasitaemia
Keywords: stepped wedge; cluster randomized controlled trial; CRCT; malaria; Plasmodium falciparum; asymptomatic carriage; mass drug administration; MDA; parasite reservoir; seasonal malaria transmission; Senegal; youth-targeted; seasonal malaria chemoprevention; SMC
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster randomized controlled trial with three steps: step 0, observation of all clusters without intervention; step 1, intervention in 50% of clusters during a year; step 2, interventions in all clusters during a year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDA and targeted control (Experimental): Interventions:
  * MDA with DHAp and SLD Primaquine
  * Targeted control (10-24 years) during the malaria high tranmission season: behaviour
  * Targeted control (15-24 years) during the malaria high tranmission season: test and treat
  During intervention period, villages receive 2 rounds of MDA simultaneously to SMC rounds 1 and 5. SMC-eligible children participate in MDA in replacement of round 1 and 5, but receive SMC rounds 2, 3 and 4 routinely.
  Youth-targeted control activities take place during the high transmission season: behavioural activies throughout and testing of asymptomatic young adults from 1 month after MDA1 to 1 month before MDA2.
  Interventions: Drug: MDA with DHAp and SLD Primaquine; Behavioral: Targeted control (10-24 years) during the malaria high tranmission season: behaviour; Diagnostic Test: Targeted control (15-24 years) during the malaria high tranmission season: test and treat
- Routine malaria control (No Intervention): Control arm will benefit from the routine malaria control strategy implemented by the Senegalese NMCP including:
  * universal coverage with long-lasting LLINs (renewed every 3 years);
  * free, community-based access to early diagnostic and treatment of malaria including active case detection activities by CHWs (DSDOM);
  * IPT for pregnant women using SP;
  * SMC for children aged 3 months to 10 years using SP+AQ, distributed door-to-door with 3-day DOTS, over 5 rounds (round 1: June; round 5: October)

INTERVENTIONS:
Drug: MDA with DHAp and SLD Primaquine — MDA: 2 rounds of MDA with dihydroartemisinine-piperaquine + single low dose primaquine (PQ) administered instead of SMC round 1 and 5.
  Arms: MDA and targeted control
Behavioral: Targeted control (10-24 years) during the malaria high tranmission season: behaviour — Communication and community engagement activities by age-groups:
  * children aged 10-14 and their parents : promote early health seeking behaviour in case of symptoms
  * young adults (15-24) : promote early health seeking behaviour in case of symptoms, emphasing the importance of mild symptoms.
  Arms: MDA and targeted control
Diagnostic Test: Targeted control (15-24 years) during the malaria high tranmission season: test and treat — Voluntary testing for malaria in young adults (15-24 years) using rapid diagnostic tests performed by community health workers during home visits or group testing events organized by the village youth association.
  Arms: MDA and targeted control

SUMMARY:
Strategies implemented since 2010 by the Senegalese National Malaria Control Program (NMCP) enabled a reduction of malaria transmission. However, malaria incidence increased again in recent years, especially in the "red zone" of Kedougou, Kolda and Tambacounda regions. Neighbouring Sahelian countries also documented an increase in malaria incidence in the same period. Current interventions include : long-lasting insecticidal nets, free diagnostic and treatment of clinical malaria, home-based case management (PECADOM), intermittent preventive treatment of pregnant women and seasonal malaria chemoprevention for children up to 10 years. These strategies, while efficient to reduce the burden of clinical malaria, do not account for individuals chronically infected with Plasmodium parasites. These carriers often remain asymptomatic and act as a reservoir for persistence during the dry season, and onwards transmission during the wet season. An observational study conducted in Kedougou in 2021 and 2022 by IRD Dakar shed light on the most affected age groups and on risk-factors associated with asymptomatic carriage.

Interventions against asymptomatic carriage could complement existing strategies and contribute to reducing malaria transmission. Mass drug administration (MDA) involves proposing a curative treatment of each member of the community, regardless of age, during a coordinated campaign. To this day, it is the only intervention available to deplete the reservoir of Plasmodium carriers, since a large proportion of asymptomatic infections remain undetectable with available field tests. A study conducted by NMCP and Iba Der Thiam University in Thiès (UIDT) in 2021 in Tambacounda showed that regular MDA campaigns during the high transmission season had a significant impact on clinical malaria incidence and on prevalence of carriage.

AMARETi project aims to evaluate an intervention to complete current control strategies. The design of this intervention combines the recent results from Kedougou and Tambacounda studies. The intervention consists of an MDA campaign at the start and at the end of the high transmission season, aiming at maximal depletion of the asymptomatic reservoir, and of age-group targeted interventions aiming to reduce chronic reinfection in individuals at highest risk of asymptomatic carriage.

The design and implementation of the intervention stem from a co-construction process with members of communities participating in the research, to maximize inclusiveness and adhesion. It aims to ensure the design of interventions that are adapted to age, gender and other factors deemed relevant by researchers and communities.

The project will evaluate if this intervention improves significantly the situation compared to current strategy in a stepped-wedge cluster-randomized controlled trial over 2 malaria high transmission seasons. If the results are conclusive, recommendations for scale-up can be made. The primary outcome will be Plasmodium falciparum infection prevalence at the end of the high transmission season. Secondary outcomes include clinical malaria incidence and malaria incidence dynamics, as well as participation, safety and acceptability.

Implementation outcomes (not detailed here) will include the assessment of implementation (CFIR's indicators), sustainability (Schell's indicators) and scalability (Coroa's indicators). These indicators use multiple dimensions stemming from qualitative and quantitative data and flexible design to understand each specific outcome (Proctor E, et al, Mental Health and Mental Health Services Research 2011).

In addition, a nested study in 10 villages will provide insights on transmission and reservoir restoration mechanisms through follow-up of a cohort and in-depth investigations.

AMARETi project will take place from 2024 to 2027 in 7 health posts and 50 villages of Kedougou department, under the leadership of the Kedougou Health District and Region authorities. The local health, administrative and community-based authorities at local and regional level are also key partners in the project, as well as local development committees and health community-based organisations. Healthpost staff and community health workers and volunteers will be essential for the operational field implementation.

ELIGIBILITY:
Randomisation unit : cluster, defined as village or group of eligible villages <3km from each other

VILLAGE-LEVEL CRITERIA Inclusion

* in Kedougou health district
* population <1500 inhabitants
* >5km from international border
* >3km from a town with 1500 inhabitants or higher
* >3km from another village/cluster

Exclusion

* village inaccessible during rainy season
* village without community health worker and impossible to set up one

INDIVIDUAL-LEVEL: MDA with DHA-piperaquine and single low dose primaquine Inclusion

* consent (+ assent for youth aged 12-17)
* age >=3 months
* in the village for >=4 days at time of MDA initiation
* not pregnant (women 15-49 years with negative pregnancy test or under contraception)

Exclusion (excluded from DHA-piperaquine and primaquine)

* allergy to artemisinin combination therapy
* pregnant women (referred for administration of IPTp) or women without pregnancy test result
* presenting with acute disease symptoms: in case of fever or history of fever, individuals will be tested with RDT and, if positive, refered to CHW or healthpost for symptomatic malaria treatment according to national guidelines.

Exclusion (excluded from primaquine only, eligible for DHA-p)

* children aged 3-6 months
* lactating women

INDIVIDUAL-LEVEL: youth-targeted testing and treatment activity Inclusion

* age 15-24 (+ assent for youth aged 15-17)
* consent Exclusion
* none. in case of RDT-positivity, participants will be referred for treatment according to national guidelines (recommendation of treatment in case of a positive test, irrespective of symptoms).

COHORT STUDY 8 villages/clusters selected for an in-depth cohort study

Household inclusion

* consent of head of household
* not planning to move out of study village
* 50% of more members aged >=15 years agree to participate

Individual participant inclusion

* household member or visitor staying longer than 1 night
* consent (+ assent for youth aged 12-17)
* age >=6 months

Individual participant exclusion

* in another study on malaria or health

Ages: 3 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18000 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Plasmodium falciparum carriage reservoir at the end of the high transmission season (step 0) | 4 months after SMC round 1, baseline year 0
  Number of participants with P. falciparum infection (measured by qPCR in cross sectional sample). Survey conducted at step 0 (baseline, year 0, no intervention). Survey takes place 4 months after SMC round 1 i.e. immediately before SMC round 5.
Plasmodium falciparum carriage reservoir at the end of the high transmission season (step 1) | 4 months after MDA1/SMC round 1, year 1
  Number of participants with P. falciparum infection (measured by qPCR in cross sectional sample). Surveys conducted at step 1 (year 1, intervention in 50% of clusters). Survey takes place 4 months after SMC round 1 in control villages (i.e. immediately before SMC round 5) and 4 months after MDA1 in intervention villages (i.e. immediately before MDA2).
Plasmodium falciparum carriage reservoir at the end of the high transmission season (step 2) | 4 months after MDA3, year 2
  Number of participants with P. falciparum infection (measured by qPCR in cross sectional sample). Surveys conducted at step 2 (year 2). During the final step, intervention MDA3 (at the start of the wet season, replacing SMC round 1) and MDA4 (at the end of the wet season, replacing SMC round 5) take place in all clusters. Survey takes place 4 months after MDA3 in intervention villages (i.e. immediately before MDA4).
Odds ratio of P. falciparum infection associated with intervention/control period status | 4 months after SMC round 1, years 0, 1 and 2
  The results of the cross sectional surveys at year 0, 1 and 2 (see outcomes 1-3) will be analysed in a multivariable multilevel logistic regression model. Explained variable : P. falciparum infection detected by qPCR. Variable of interest : intervention or control status at village level. Adjustments for individual, household, and cluster-level fixed effects. Including household, village, cluster and temporal random effects.

SECONDARY OUTCOMES:
Clinical malaria burden | year 1, year 2
  Cumulative P. falciparum clinical malaria incidence in study villages during the high transmission season (june to january) as recorded at community (CHW) and health-facility level. Comparison between intervention and control periods will evaluate burden reduction associated with intervention status.
Spatio-temporal dynamics of clinical malaria incidence | year 1, year 2
  Time-series of weekly cumulative incidence of clinical P. falciparum malaria recorded by CHW and health facilities in study villages during the high transmission season.
Mass drug administration safety (active) | Day 4 after MDA start
  Frequency and severity of adverse events identified by active detection in a random sample of participants immediately after each MDA round.
Mass drug administration safety (passive) | Day 0 to day 7 after MDA start
  Frequency and severity of adverse events recorded by passive detection at community (CHW) and health-facility level during each MDA (MDA1, 2, 3 and 4).
Plasmodium falciparum carriage reservoir at the onset of the high transmission season (step 1) | immediately before MDA1/SMC round 1, year 1
  Number of participants with P. falciparum infection (measured by qPCR in cross sectional sample). Survey conducted at step 1 (year 1, intervention in 50% of clusters). Survey takes place immediately before SMC round 1 in control villages and immediately before MDA1 in intervention villages. This period corresponds to the onset of the high transmission season (i.e. the end of the dry, low transmission season)
Plasmodium falciparum carriage reservoir at the onset of the high transmission season (step 2) | immediately before MDA3, year 2
  Number of participants with P. falciparum infection (measured by qPCR in cross sectional sample). Surveys conducted at step 2 (year 2, intervention in 100% of clusters), immediately before MDA3, at the onset of the high transmission season (i.e. at the end of the dry, low transmission season)
Plasmodium falciparum infection prevalence in 10-14 and 15-24 years | 4 months after SMC round 1 / MDA1, year 1
  Number of participants aged 10-14 and 15-24 years with P. falciparum infection (measured by qPCR in cross sectional sample). Surveys conducted at step 1 (year 1, intervention in 50% of clusters). Survey takes place 4 months after SMC round 1 in control villages (i.e. immediately before SMC round 5) and 4 months after MDA1 in intervention villages (i.e. immediately before MDA2). This subgroup analysis of secondary outcome 2 will enable comparison of prevalence and prevalence reduction between intervention and control periods by age-group to estimate potential effectiveness of the targeted control intervention.
Plasmodium falciparum infection prevalence in 10-14 and 15-24 years | 4 months after MDA3, year 2
  Number of participants aged 10-14 and 15-24 years with P. falciparum infection (measured by qPCR in cross sectional sample). Surveys conducted at step 2 (year 2, intervention in all clusters). Survey takes place 4 months after MDA3 (i.e. immediately before MDA4). This subgroup analysis of secondary outcome 3 will enable comparison of prevalence and prevalence reduction between intervention and control periods by age-group to estimate potential effectiveness of the targeted control intervention.
Intervention cost-effectiveness | year 2 and year 3
  Intervention cost and cost-effectiveness ratio regarding prevalence reduction and clinical burden reduction
Participation to MDA intervention | Day 5 after MDA (MDA1 & MDA2, year 1; MDA2 & MDA3, year 2).
  Proportion of population participating to intervention relatively to total and eligible population, estimated for each MDA round (MDA1 to MDA4). 3-dose complete participation measured at the end of each MDA round, as well as incomplete participation (only 1 or 2 doses taken).
Participation to targeted control intervention (15-24 years) | from month 2 to month 3 MDA1 (year 2) ; from month 2 to month 3 after MDA3 (year 2)
  Proportion of eligible 15-24 years old who completed at least one rapid diagnostic test during targeted control activities taking place from month 2 to month 3 after MDA1 during year 1 and from month 2 to month 3 after MDA3 during year 2.
Intervention acceptability | after MDA, year 1
  Sekhon's indicators of acceptability evaluated using mixed methods (quantitative during cross-sectional surveys and qualitative) evaluated prospectively before MDA and retrospectively after MDA. Quantitative evaluation will rely on a -7 to +7 scale established combining responses to close-ended questions on the 7 dimensions of acceptability.

OTHER OUTCOMES:
Risk-factors for Plasmodium falciparum infection in a subcohort follow-up | 6 planned cohort visits (from baseline year 0 to 4 months after MDA3, during year 2).
  Plasmodium falciparum qPCR positivity odds-ratio in a multivariable multilevel logistic regression model including fixed effects (age, sex and relevant exposure covariables) and spatial and temporal random effects at individual, household, village, cluster and period levels. This analysis includes 6 cohort visits :
  1. baseline at 4 months after SMC1 during year 0;
  2. immediately before SMC1/MDA1 during year 1;
  3. 2 months after SMC1/MDA1 during year 1;
  4. 4 months after SMC1/MDA1 during year 1;
  5. immediately MDA3 during year 2;
  6. 4 months after MDA3 during year 2.
Subcohort villages parasite reservoir genetic relatedness | year 1, year 2
  Genetic relatedness (identity by descent) between Plasmodium parasites genotyped after detection in individuals presenting symptomatic, Rapid Diagnostic Test-confirmed P. falciparum malaria episodes during the high transmission season or in P. falciparum infected participants in surveys (see primary outcome and secondary outcome 9 and 10).
Subcohort villages parasite reservoir multiplicity of infection | year 1, year 2
  Multiplicity of infection quantified after Plasmodium parasite genotyping in individuals presenting symptomatic, Rapid Diagnostic Test-confirmed P. falciparum malaria episodes during the high transmission season or in P. falciparum infected participants in surveys (see primary outcome and secondary outcome 9 and 10).
Rapid Diagnostic Test positivity rate in youths (15-24 years) participating to targeted control testing activity | Month 2 and Month 3 after MDA1 (step 1) or MDA3 (step 2)
  Intervention arm only: evaluate the number and frequency detection to estimate the potential impact on the reservoir.

CONTACTS AND LOCATIONS:
Locations (1):
- District de Santé de Kédougou - Kedougou Health District, Kédougou, Senegal

IPD SHARING:
Plan to Share IPD: Undecided